CLINICAL TRIAL: NCT06683300
Title: Drug Eluting Stenting and Short Dual Antiplatelet Therapy for Preventing Recurrent Stroke in Vertebral Stenosis Registry Study
Acronym: M Short DAPT
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024-158-02
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Vertebral Artery Stenosis
Keywords: vertebral artery stent; dual antiplatelet duration; symptomatic vertebral artery atherosclerotic stenosis
MeSH Terms: conditions — Vertebrobasilar Insufficiency | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 3 months DAPT: dual antiplatelet therapy (DAPT) for 3 months
  Interventions: Drug: DAPT for 3 months after vertebral artery stenting

INTERVENTIONS:
Drug: DAPT for 3 months after vertebral artery stenting — After implantation of a drug-eluting stent in the vertebral artery, dual antiplatelet therapy (DAPT) were administered for 3 months. The types of antiplatelet medications are not limited, with the standard regimen consisting of aspirin 100 mg once daily combined with either clopidogrel 75 mg once daily or ticagrelor 90 mg twice daily. Additional antiplatelet agents such as indobufen may also be considered acceptable.

SUMMARY:
This is a prospective, multi-center, registry study exploring the duration of dual antiplatelet therapy (DAPT) after drug-eluting stent(DES) treatment of symptomatic vertebral artery atherosclerotic stenosis. The trial will be conducted in approximately 30 interventional neurology centers in China.

Currently, there is no consensus regarding the duration of DAPT after drug-eluting stent treatment for vertebral artery stenosis(VAS). The objective of this study is to standardize clinical medication by shortening the duration of DAPT, thereby reducing the bleeding risk and medication burden for patients, while ensuring that there is no increase in ischemic events.

DETAILED DESCRIPTION:
As the drug-eluting stents (DES) with indications for vertebral artery treatment have been officially approved in China, DES has gradually been widely used in the treatment of vertebral artery stenosis. There is increasing clinical attention towards the duration of dual antiplatelet therapy (DAPT) following stenting.

Currently, there is limited evidence regarding the optimal DAPT duration following endovascular treatment for vertebral artery stenosis. Therefore, clinical practice typically relies on experiences derived from treatments for coronary, carotid, or lower limb artery diseases, with a conventional recommendation of 6 to 12 months of antiplatelet therapy post-stent implantation.

Evidence obtained from coronary stents shows that the short-term DAPT strategy of 1-3 months after PCI in the new generation of DES can significantly reduce the incidence of severe bleeding without increasing ischemic events compared with the standard DAPT strategy of 7-12 months, especially for non-acute elective surgery patients who are similar to those with vertebral artery stenosis stents.

This study employs new-generation Co-Cr fluoropolymer DES to evaluate the balance between ischemic and bleeding complications by shortening the DAPT duration, with the ultimate aim of maximizing patient benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender unlimited;
2. Based on clinical and imaging evidence, the investigators identified patients with symptomatic vertebral atherosclerotic stenosis who met the indications for the placement of drug-eluting vertebral artery stents;
3. Patients or their guardians sign informed consent.

Exclusion Criteria:

1. Severe coagulation dysfunction, serious uncontrolled infection, serious systemic disease, uncontrolled hypertension, etc., are not suitable for surgery;
2. Patients with aneurysms that cannot be treated in advance or at the same time or are not suitable for surgery;
3. Myocardial infarction or large-scale cerebral infarction occurred within 2 weeks;
4. Combined with atrial fibrillation, or accompanied by serious heart, liver, kidney and lung diseases;
5. Interventional or surgical procedures are planned within 90 days;
6. Known contraindications to heparin, rapamycin, anesthesia and contrast agents;
7. Life expectancy is less than 12 months;
8. The researcher considers it inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic vertebral atherosclerotic stenosis who met the indications for the placement of drug-eluting vertebral artery stents.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ischemic stroke in the territory of the target artery within 1 year | 12 months after stent implantation
  The primary endpoint was defined as occurrence of ischemic stroke events in the target arterial territory, excluding transient ischemic attacks.

SECONDARY OUTCOMES:
Occurrence of Periprocedural events | within 30 days after stent implantation
  Periprocedural events defined as occurrence of transient ischemic attack (TIA), ischemic stroke and all-cause death.
Occurrence of Bleeding Events within 1 year | 12 months after stent implantation
  Bleeding events are defined as gastrointestinal hemorrhage, gingival hemorrhage, conjunctival hemorrhage, intraocular hemorrhage, nasal hemorrhage, hemoptysis, cerebral hemorrhage(such as subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH), or subdural hematoma (SDH)), bleeding at puncture sites, intraperitoneal bleeding, and skin bleeding, among others.
Occurrence of TIA events related to the target territory within 1 year | 12 months after stent implantation
  The outcome defined as temporary neurological symptoms caused by TIA that related to the target lesion judged by physicians.
Occurrence of disabling and fatal stroke events within 1 year | 12 months after stent implantation
  Disabling and fatal stroke are defined as stroke that results in severe disability or death.
AEs and SAEs | in 12 months
Occurrence of residual stenosis after the procedure | At the end of the procedure
  Degree of residual stenosis was measured and calculated according to the methods of the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) trial.
Rate of In-stent restenosis (ISR) within 12 months | 12 months after stent implantation
  The ISR is defined as >50% stenosis within or immediately adjacent (within 5 mm) of the implanted stent and >20% absolute luminal loss.
modified Rankin Scale score at 1 year | 12 months after stent implantation
  The range of modified Rankin Scale was from 0 to 6. 0-No symptoms;
  1. No significant disability;
  2. Slight disability;
  3. Moderate disability;
  4. Moderately severe disability;
  5. Severe disability; 6 -Dead. A higher score indicates a poorer outcome.
The National Institutes of Health Stroke Scale (NIHSS) score at 1 year | 12 months after stent implantation
  NIHSS is a standardized scoring system used to measure the severity of neurological deficits caused by a stroke. It assesses various aspects of brain function, including consciousness, vision, sensation, movement, speech, and language. The scale ranges from 0 to 42, with higher scores indicating more severe strokes.
EQ-5D score at 1 year | 12 months after stent implantation
  The EQ-5D is a standardized questionnaire used to measure health-related quality of life. It assesses five dimensions of health: Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression. Each dimension is scored from 1 to 3, with 1 being no problems, 2 being some or moderate problems, and 3 being severe or extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes